CLINICAL TRIAL: NCT02626702
Title: Immune Modulators in Women Undergoing IVF----a Prospective Study
Brief Title: Immune Modulators and IVF
Status: Terminated | Type: Observational
Why Stopped: Lab close down
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1502015953
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: In Vitro Fertilization
Keywords: immune modulators; IVF outcomes; relationship
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Excess blood from subjects will be analyzed to explore the relationship between Immune Modulators and IVF outcomes.

SUMMARY:
Exploring the immune mediators of early pregnancy prospectively may help to identify new early interventions that will increase the likelihood of success and help women make informed decisions regarding their pregnancies.

DETAILED DESCRIPTION:
Sera will be obtained from 500 women undergoing IVF at five time periods: cycle Day 2, post HCG, Day 24, Day 28, and/or Day 35.Aliquots of sera will be tested by commercial ELISA kits for concentrations of immune modulators suggestive to be predictive of IVF outcome, such as cytokines (interleukins, tumor necrosis factor, and interferon), neurotrophins (BDNF), protease inhibitors (HE4) and insulin-like growth factors (IGF-1, IGF-2, IGFBP). The results will be correlated with IVF outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All fresh transfers

Exclusion Criteria:

* PGD

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects undergoing In Vitro Fertilization.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-07-31; Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
To explore the relationship between immune mediators and IVF outcome prospectively in women who receive in vitro fertilization treatment. | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Spandorfer, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Ronald O. Perelman and Claudia Cohen Center for Reproductive Medicine, New York, New York, United States